CLINICAL TRIAL: NCT00564915
Title: RCT of the Efficacy of the Ketogenic Diet in the Treatment of Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Child Health (Other)
Responsible Party: Tracy Assari, Institute of Child Health
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 98NR04
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Epilepsy
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — Ketogenic diet

SUMMARY:
A study of the efficacy and tolerability of two different ketogenic diets in children with drug resistant epilepsy; children resistant to at least two drugs randomised to reveive diet after baseline or after further 3m control period; in addition randomised to either MCT or classical ketogenic diet.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy for at least 2 years, resistant to at least two AEDs, at least 7 seizures/week

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2001-12; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Change in seizure frequency | 3 months

SECONDARY OUTCOMES:
Tolerability and assessment of ketosis and growth | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Helen Cross, Professor, Principal Investigator — UCL Institute of Child Health
Locations (1):
- Institute of Child Health, The Wolfson Centre, London, United Kingdom

REFERENCES:
- [Derived] Neal EG, Chaffe H, Schwartz RH, Lawson MS, Edwards N, Fitzsimmons G, Whitney A, Cross JH. The ketogenic diet for the treatment of childhood epilepsy: a randomised controlled trial. Lancet Neurol. 2008 Jun;7(6):500-6. doi: 10.1016/S1474-4422(08)70092-9. Epub 2008 May 2. PMID 18456557